CLINICAL TRIAL: NCT05361005
Title: A Phase Ic Single Center, Randomized, Double-Blind, Placebo-controlled, Single Dose Escalation and Multiple Dose Study to Evaluate the Tolerability and Pharmacokinetics of BDB-001 Injection in Healthy Subjects
Brief Title: Tolerability and Safety of BDB-001 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Beijing Defengrei Biotechnology Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STS-BDB001-05
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — BDB001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 2mg/kg (Experimental): All participants (fasted) received either 2 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 4mg/kg (Experimental): All participants (fasted) received either 4 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 8mg/kg (Experimental): All participants (fasted) received either 8mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 4mg/kg multiple doses (Experimental): All participants (fasted) received either 4 mg/kg of BDB-001 as a multiple doses or doses-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo

INTERVENTIONS:
Drug: BDB-001 injection — Intravenous injection
Drug: Placebo — Intravenous injection

SUMMARY:
A clinical study to evaluate the tolerability, PK and PD characteristics of BDB-001 Injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18~55 years old (including 18 and 55 years old);
* A healthy subject evaluated by medical history etc;
* Physical examination and vital signs normal, or abnormal without clinical significance;
* Weight: 80 kg ≥ male ≥50 kg, and 80 kg ≥ female ≥45 kg. Body Mass Index (BMI) between 18~28kg/m2 (including 18 and 28). Body mass index (BMI) = body weight (kg) / height 2 (m2);
* Be able to complete the study in compliance with protocol;
* The subjects (including sex partners) willing to take effective contraception measures within 6 months after the last dose. Refer to the appendix for the detailed contraceptive methods;
* Informed consent form signed prior to the study and the content, process and possible adverse reactions of the study fully understood.

Exclusion Criteria:

* More than 5 cigarettes were smoked daily within 3 months prior to screening period of the study;
* Allergic history (drugs and food);
* A history of drug abuse and / or drinking (drinking 14 units per week of alcohol: 1 unit = 285 mL beer, or liquor 25 mL, or wine 100ml);
* Subjects who had donated blood or massive blood loss (> 450 mL) within 3 months prior to screening period, or those who had plasma exchange within 4 weeks prior to screening period;
* Any prescription drugs, OTC drugs, any vitamin products or herbs were used within the 14 days prior to screening period, and immunomodulators were used within 28 days prior to screening period;
* Subjects who had taken other investigational product(s) or vaccine within 3 months prior to screening period, or those who were expected to be vaccinated within 2 months after completion of the study;
* Vigorous exercise or other factors affecting drug absorption, distribution, metabolism, excretion within 2 weeks prior to screening;
* Significant change in eating or exercise habits recently;
* Subjects who have taken BDB-001 injection or participated in clinical trials of investigational drugs within three months prior to taking study drugs;
* Subjects with a history of previous tuberculosis and exposure to active tuberculosis, TB-spot test results is greater than 2 UL(upper limit) of normal range, and those with infectious diseases recently;
* Subjects with autoimmune or immunodeficiency diseases, or with a family history of autoimmune diseases or immunodeficiency diseases;
* Abnormal ECG with clinical significance;
* Female subjects are in the lactation period or have positive serum pregnancy results during the period of trial (from screening to completion);
* Clinical laboratory examination result with clinical significance, or other clinical findings within 12 months prior to screening period with clinical significance ( including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular diseases);
* Subjects whose white blood cell count, high-sensitivity C-reactive protein test results were abnormal with clinical significance during screening and baseline period (-1 day), hemoglobin: male <120g/L or female <110g/L;
* Subjects with positive result of viral hepatitis (including hepatitis B and C), AIDS antibody, or treponema pallidum antibody;
* Subjects with acute disease or with concomitant medication from the screening stage to the start time of drug administration;
* Subjects with more than 5 cups (150mL cups) of coffee, tea or cola each day;
* Subjects with any alcohol-containing products within 48 hours before taking study medication;
* Subjects with a positive urine drug screening or with a history of drug abuse or drug use within the past five years;
* The investigators suggested the subject was not suitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities And Clinically Significant Physical Examination Abnormalities | Up to 28 Days
Maximum plasma concentration (Cmax) | Up to 504 hours postdose
Area under the plasma concentration-time curve from time 0 to infinity (AUC0inf) | Up to 504 hours postdose
Area under the plasma concentration-time curve from time 0 to 480hr(AUC00-480hr) | Up to 504 hours postdose
Time of maximum concentration (Tmax) | Up to 504 hours postdose
Elimination half-life (t1/2) | Up to 504 hours postdose
Clearance (CL) | Up to 504 hours postdose
Apparent volume of distribution (Vz) | Up to 504 hours postdose
Mean residence time (MRT) | Up to 504 hours postdose

SECONDARY OUTCOMES:
Change from baseline in concentration of free C5a and anti-drug antibody | Up to 504 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Shu Lan (Hangzhou) Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No